CLINICAL TRIAL: NCT02257073
Title: Cognitive-behavioral Treatment for Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Dr., Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBRA20140102; BWS11J067 (Other Grant/Funding Number: "Twelfth Five-Year Plan" Scientific Research Funds Project of Chinese PLA)
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT (Experimental): Cognitive-behavioral treatment
  Interventions: Behavioral: Cognitive-behavioral treatment
- WLT (Sham Comparator): Waiting in list
  Interventions: Behavioral: Waiting List

INTERVENTIONS:
Behavioral: Cognitive-behavioral treatment
  Arms: CBT
Behavioral: Waiting List
  Arms: WLT

SUMMARY:
To evaluate the effectiveness of Cognitive-behavioral treatment for people with rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by rheumatology consultants with RA

Exclusion Criteria:

* severe psychological difficulties
* currently receiving mental health care
* any medical condition that might prevent them from safely exercising (e.g. history of more severe heart, lung or cerebrovascular disease)
* previously attended an education programme
* had a Modified Health Assessment Questionnaire score >2 (score range 0-3), that is severe functional problems
* history of organic brain syndrome
* presence of a psychotic disorder
* presence of other uncontrolled medical disorders
* presence of a major communication disorder, illiteracy
* presence of less than an 8th grade education (due to inability to complete questionnaires)
* presence of a therapeutic dosage of an antidepressant medication, or presence of another autoimmune disease/disabling condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in disease activity score in 28 joints(DAS28) at 48 weeks | at 0 week, 12 weeks, 24 weeks, 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chengdu Military Area Command PLA, Chengdu, Sichuan, China